CLINICAL TRIAL: NCT03451045
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 2 Trial to Evaluate Efficacy and Safety of Lenabasum in Cystic Fibrosis
Brief Title: Trial to Evaluate Efficacy and Safety of Lenabasum in Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corbus Pharmaceuticals Inc. (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JBT101-CF-002
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Cystic Fibrosis
Keywords: Pulmonary exacerbation, lenabasum, JBT-101
MeSH Terms: conditions — Cystic Fibrosis | interventions — lenabasum

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind, randomized, placebo-controlled, parallel group study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lenabasum 20 mg BID (Experimental)
  Interventions: Drug: Lenabasum 20 mg
- Lenabasum 5 mg BID (Experimental)
  Interventions: Drug: Lenabasum 5 mg
- Placebo BID (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lenabasum 20 mg — Subjects will receive lenabasum 20 mg twice daily.
  Arms: Lenabasum 20 mg BID
Drug: Lenabasum 5 mg — Subjects will receive lenabasum 5 mg twice daily.
  Arms: Lenabasum 5 mg BID
Other: Placebo — Subjects will receive placebo twice daily.
  Arms: Placebo BID

SUMMARY:
This is a Phase 2 multicenter, double-blind, randomized, placebo-controlled study assessing the efficacy and safety of lenabasum for the treatment of cystic fibrosis in patients 12 years of age or older. Approximately 415 subjects will be enrolled in this study at about 100 sites in North America, and Europe. The planned duration of treatment with study drug is 28 weeks.

Study drug will be lenabasum 20 mg BID, lenabasum 5 mg BID, and placebo in a 2:1:2 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 12 years of age at the time Informed Consent/ Assent is signed.
2. Weight ≥ 40 kg.
3. FEV1 ≥ 40% predicted and < 100% predicted in the last 12 months.
4. Physician-initiated treatment with an IV antibiotic 2 or 3 times in the last 12 months for a new PEx or physician-initiated treatment with an IV antibiotic 1 time in the last 12 months plus physician-initiated treatment with oral antibiotic(s) 1 or more times in the past 12 months for a new PEX.

Exclusion Criteria:

1. Severe or unstable CF at screening or Visit 1.
2. Any of the following values for laboratory tests at screening:

   1. A positive pregnancy test.
   2. Hemoglobin < 10 g/dL in males and < 9 g/dL in females.
   3. Neutrophils < 1.0 x 10^9 /L.
   4. Platelets < 75 x 10^9/L.
   5. Creatinine clearance < 50 mL/min according to Modification of Diet in Renal Disease (MDRD) Study equation.
   6. Serum transaminases > 2.5 x upper limit of normal.
3. Any medical condition or concurrent medical therapies at screening or Visit 1 that may put the subject at greater safety risk, influence response to study drug or interfere with study assessments.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Chmiel, MD, Principal Investigator — Indiana University School of Medicine/Riley Physicians Pulmonary; J. Stuart Elborn, MD, Principal Investigator — National Heart and Lung Institute, Imperial College
Locations (105):
- United States (34):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Miller Children's Hospital, Long Beach, California
  - National Jewish Health, Denver, Colorado
  - University of Miami, Miami, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - USF Center for Advance Lung Disease, Tampa, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The Cystic Fibrosis Institute, Glenview, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center (main location), Lebanon, New Hampshire
  - Dartmouth-Hitchcock Manchester (satellite site), Manchester, New Hampshire
  - Atlantic Health Children's Hospital, Morristown, New Jersey
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - New York Medical College, Hawthorne, New York
  - North Shore LIJ Health System, New Hyde Park, New York
  - Mount Sinai Beth Israel, New York, New York
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Milton S. Hershey Medical Center / Penn State College of Medicine, Hershey, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Children's Specialty Clinic, Sioux Falls, South Dakota
  - UT Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - University Hospital and UW Health Clinics, Madison, Wisconsin
- Austria (2):
  - Cystic Fibrosis Centre Innsbruck Medical University of Innsbruck, Dept. for Child and Adolescent Health, University Clinic for Paediatrics, Cardiology, Pneumology, Allergology, Cystic Fibrosis, Innsbruck
  - Medical University of Vienna, Vienna
- Universitair Ziekenhuis Brussel, Brussels, Belgium
- Bulgaria (3):
  - Medical Center Prolet EOOD, Rousse
  - UMHAT Alexandrovska, Sofia
  - MHAT Sveta Marina EAD, Varna
- Canada (4):
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal
  - St. Michael's Hospital, Toronto
  - The Hospital for Sick Children, Toronto
  - St. Paul's Hospital, Vancouver
- Motol University Hospital, Prague, Czechia
- France (10):
  - Centre de Référence de la Mucoviscidose, Bron
  - Service de Pneumologie, Allergologie, Mucoviscidose; Hôpital Femme-Mère-Enfant, Bron
  - Service de Pediatrie Medico-Chirurgicale et Genetique, Dijon
  - CHRU de Montpellier, Montpellier
  - CRCM Enfant de Nancy, Nancy
  - CHU de Nice, Nice
  - Centre de Recherche en Explorations Fonctionnelles (CREF), Paris
  - CRCM Hôpital Necker, Paris
  - Foundation ILDYS, Roscoff
  - Nouvel Hopital Civil Strasbourg, Strasbourg
- Germany (8):
  - Charité Universitätsmedzin, Berlin
  - Catholic Hospital Bochum - St. Josef-Hospital, Bochum
  - University Hospital Essen, Essen
  - University Medicine Essen Ruhrlandklinik, Essen
  - Goethe University Children´s Hospital, Frankfurt
  - Hannover Medical School, Hanover
  - University Hospital Jena, Jena
  - Klinikum der Ludwig Maximilian Universität München, München
- General Hospital of Thessaloniki Ippokratio, Thessaloniki, Greece
- Hungary (5):
  - National Koranyi Institute of Pulmonology, Department of Cystic Fibrosis, Budapest
  - University of Debrecen - Kenezy Gyula University Hospital, Debrecen
  - Bács-Kiskun County Hospital, Teaching Hospital of the University of Szeged, Kecskemét
  - Moritz Kaposi General Hospital, Mosdós, Department of Pediatric Pulmonary Rehabilitation, Mosdós
  - Pediatric Pulmonology, Törökbálint, Hungary, Törökbálint
- Italy (5):
  - Centro Regionale Toscano di Riferimento per la Fibrosi Cistica, Florence
  - U.O.S.D. - Centro fibrosi cistica, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Verona, Verona
- Radbound UMC, Nijmegen, Netherlands
- Poland (4):
  - Instytut Matki I Dziecka, Centrum Leczenia Mukowiscydozy - Oddzial Chorob Pluc, Dziekanów Leśny
  - Oddzial Pediatrii z Pododdzialem Leczenia Mukowiscydozy, Gdansk
  - Instytut Gruzlicy I Chorob Pluc Oddzial Terenowy im Jana I Ireny Rudnikow, Rabka-Zdrój
  - Institute for Mother and Child, Department of CF for Children's and Youth, Rzeszów
- Hospital de Santa Maria, Lisbon, Portugal
- Medial Center for Ambulatory Diagnosis and Treatment, Brasov, Romania
- Russia (4):
  - Scientfic Research Institute of Pulmonology, Moscow
  - Diagnostic Children Hospital, Department of Pediatrics and Adolescent Medicine, Department of Pediatric Pulmonary, Allergology and Endocrinology, Mytishchi
  - Children's City Hospital of Saint Olga, Saint Petersburg
  - First St. Petersburg State Pavlov Medical University, Saint Petersburg
- Serbia (3):
  - Clinical for Pulmonary Diseases, Clinical Center of Serbia, Belgrade
  - Institute for Pulmonary Disease of Vojvodina, Kamenitz
  - Institute for Child and Youth Health Care of Vojvodina, Novi Sad
- Slovakia (2):
  - Children's faculty hospital with polyclinic Banska Bystrica, Banská Bystrica
  - Children's Faculty Hospital Kosice, Košice
- Spain (3):
  - Unidad de Fibrosis Quistica Adultos, Barcelona
  - Unidad de Fibrosis Quistica Pediatria, Barcelona
  - Unidad de Fibrosis Quistica y Transplante Pulmonar, Valencia
- Sweden (2):
  - Skane University Hospital, Lund
  - Karolinska University Hospital, Stockholm
- United Kingdom (10):
  - Liverpool Heart and Chest Hospital, Liverpool, Merseyside
  - Belfast City Hospital, Belfast, Northern Ireland
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Cardiff and Vale University Health Board, Llandough
  - Barts Health NHS Trust, London
  - Royal Brompton & Harefield NHS Foundation Trust, London
  - Wolfson Cystic Fibrosis Centre City Hospital Campus, Nottingham
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: subjects received placebo BID
Period: Overall Study
Arm/Group | Lenabasum 20 mg BID | Lenabasum 5 mg BID | Placebo
Started | 175 | 91 | 181
Completed | 148 | 85 | 154
Not Completed | 27 | 6 | 27
Not completed — Lack of Efficacy | 3 | 2 | 2
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 0 | 5
Not completed — Pregnancy | 0 | 0 | 2
Not completed — Adverse Event | 7 | 1 | 3
Not completed — Non-compliance with study | 2 | 0 | 1
Not completed — any other reason | 10 | 2 | 13

BASELINE CHARACTERISTICS:
Population: modified intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenabasum 20 mg BID | Lenabasum 5 mg BID | Placebo | Total
Number analyzed (Participants) | 165 | 89 | 171 | 425
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (9.08) | 28.9 (11.24) | 26.6 (10.81) | 26.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 44 | 93 | 228
  Male | 74 | 45 | 78 | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 5 | 13
  Not Hispanic or Latino | 155 | 84 | 164 | 403
  Unknown or Not Reported | 5 | 2 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 3 | 5
  White | 161 | 86 | 163 | 410
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 2 | 1 | 3 | 6
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 21.07 (3.179) | 22.26 (4.164) | 21.52 (3.931) | 21.50 (3.728)
FEV1 (L) [Mean (Standard Deviation); unit: liters] | 2.10 (0.73) | 2.20 (0.77) | 2.17 (0.75) | 2.15 (0.76)
Number of Acute Pulmonary Exacerbations in Past Year [Count of Participants; unit: Participants]
  one | 1 | 0 | 1 | 2
  two | 75 | 43 | 76 | 194
  three | 63 | 30 | 69 | 162
  four | 20 | 11 | 13 | 44
  five | 6 | 4 | 10 | 20
  six or more | 0 | 1 | 2 | 3
CFTR Genotype [Count of Participants; unit: Participants]
  F508del/F508del | 83 | 34 | 74 | 191
  F508del/other | 56 | 38 | 70 | 164
  Other/other or unknown | 26 | 17 | 27 | 70
Weight [Mean (Standard Deviation); unit: kg] | 58.41 (11.567) | 62.82 (15.540) | 59.25 (13.645) | 59.67 (13.390)

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Exacerbation (PEx) Rate Over 28 Weeks
Description: Rate of PEx using the primary PEx definition with lenabasum 20 mg BID compared to placebo, during the treatment period. An primary PEx is defined on the physician's decision to treat with oral, intraveneous or inhaled antibiotics in the presence 4/12 Fuch's criteria (Change in sputum, new/increased hemoptysis, increased cough, increased dyspnea, malaise, fatigue/lethargy, Temperature greater than 38C, weight loss, sinus pain, change in sinus discharge, change in exam of chest, decrease in FEV1 of more than 10%, radiographic change). This excludes prophylactic antibiotics. A new PEx is a one that occurs at 28 days after the previous PEx.
Time Frame: 28 weeks (Baseline Day 0 to Week 28)
Population: modified intent to treat population
Measure: Number; unit: events per participant/28 weeks
Arm/Group | Lenabasum 20 mg BID | Lenabasum 5 mg BID | Placebo BID
Number analyzed (Participants) | 165 | 89 | 171
events per participant/28 weeks | 0.911 | 0.749 | 0.842

2. Secondary Outcome: Pulmonary Exacerbation (PEx) Rate
Description: Event rate of PEx using the secondary PEx definition with lenabasum 20 mg BID compared to placebo. The secondary definition of a PEx is based on the physician's diagnosis of pulmonary exacerbation and commencement of new oral, intravenous, or inhaled antibiotics. A new PEx is defined one that starts 28 or more days after the previous confirmed PEx. The PEx rate is calculated as the number of PEx/28 weeks
Time Frame: 28 weeks (Baseline Day 0 to Week 28)
Population: modified intent to treat population
Measure: Number; unit: events per participant/28 weeks
Arm/Group | Lenabasum 20 mg BID | Lenabasum 5 mg BID | Placebo
Number analyzed (Participants) | 165 | 89 | 171
events per participant/28 weeks | 1.08 | 0.91 | 1.03

3. Secondary Outcome: Time to First New Pulmonary Exacerbation (PEx)
Description: Time to first new PEx using the primary PEx definition with lenabasum 20 mg BID compared to placebo. An primary PEx is defined on the physician's decision to treat with oral, intraveneous or inhaled antibiotics in the presence 4/12 Fuch's criteria (Change in sputum, new/increased hemoptysis, increased cough, increased dyspnea, malaise, fatigue/lethargy, Temperature greater than 38C, weight loss, sinus pain, change in sinus discharge, change in exam of chest, decrease in FEV1 of more than 10%, radiographic change). This excludes prophylactic antibiotics. A new PEx is a one that occurs at 28 days after the previous PEx. The rate is calculate over a 28 week period from visit 1 to week 28 visit
Time Frame: 28 weeks (Baseline Day 0 to Week 28)
Population: modified intent to treat population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lenabasum 20 mg BID | Lenabasum 5 mg BID | Placebo
Number analyzed (Participants) | 165 | 89 | 171
days | 162 [59 to 183] | 148 [58 to 183] | 143 [58 to 183]

4. Secondary Outcome: Pulmonary Exacerbation (PEx)
Description: Time to first PEx using the secondary PEx definition with lenabasum 20 mg BID compared to placebo. The secondary definition of a PEx is based on the physician's diagnosis of pulmonary exacerbation and commencement of new oral, intravenous, or inhaled antibiotics. A new PEx is defined one that starts 28 or more days after the previous confirmed PEx.
Time Frame: 28 weeks (Baseline Day 0 to Week 28)
Population: modified intent to treat population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lenabasum 20 mg BID | Lenabasum 5 mg BID | Placebo
Number analyzed (Participants) | 165 | 89 | 171
days | 116 [38 to 183] | 113 [54 to 183] | 120 [49 to 183]

5. Secondary Outcome: CFQ-R Respiratory Symptom Domain
Description: Cystic Fibrosis Questionnaire - Revised measures change from baseline in CFQ-R respiratory symptom domain with lenabasum compared to placebo. Subjects >/= 14 years of age. 5 distinct 4-point Likert scales (e.g., always/often/ sometime/never) Scores for each HRQoL domain; after recoding, each item is summed to generate a domain score and standardized. Scores range from 0 to 100, with higher scores indicating better health.
Time Frame: 28 weeks (Change from Baseline Day 0 to Week 28)
Population: modified intent to treat population
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Lenabasum 20 mg BID | Lenabasum 5 mg BID | Placebo
Number analyzed (Participants) | 165 | 89 | 171
scores on a scale | 1.16 (1.41) | -2.92 (1.88) | -0.96 (1.41)

6. Secondary Outcome: FEV1 % Predicted
Description: Change from baseline to week 28 in Forced Expiratory Volume in 1 second (FEV1) expressed as a percentage of a normal range. A lower percentage FEV1 is indicative of decrease in lung functionality. The changes observed from baseline to week 28 for lenabasum will be compared with those observed for placebo treated participants.
Time Frame: 28 weeks (Change from Baseline Day 0 to Week 28)
Population: modified intent to treat population
Measure: Least Squares Mean (Standard Error); unit: percentage of Predicted FEV1
Arm/Group | Lenabasum 20 mg BID | Lenabasum 5 mg BID | Placebo
Number analyzed (Participants) | 165 | 89 | 171
percentage of Predicted FEV1 | 0.014 (0.025) | -0.005 (0.033) | -0.012 (0.025)

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Lenabasum 20 mg BID | Lenabasum 5 mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/165 | 0/89 | 0/171
Serious Adverse Events (participants affected / at risk) | 50/165 | 25/89 | 50/171
Other Adverse Events (participants affected / at risk) | 151/165 | 80/89 | 151/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenabasum 20 mg BID (N=165) | Lenabasum 5 mg BID (N=89) | Placebo (N=171)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Tachcardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Non-compaction cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal disease carrier (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Forced expiratory volume decreased (Investigations) | 1 (2) | 0 (0) | 2 (2)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Human rhinovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary function test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Infective pulmonary exacerbation of cystic fibrosis (Respiratory, thoracic and mediastinal disorders) | 42 (61) | 22 (29) | 41 (53)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenabasum 20 mg BID (N=165) | Lenabasum 5 mg BID (N=89) | Placebo (N=171)
Gastrointestinal disorders (Gastrointestinal disorders) | 45 (79) | 23 (53) | 43 (80)
General disorders and administration site conditions (General disorders) | 39 (70) | 22 (33) | 33 (41)
Immune system disorders (Immune system disorders) | 2 (6) | 3 (4) | 5 (7)
Infections and infestations (Infections and infestations) | 75 (112) | 36 (54) | 72 (114)
Investigations (Investigations) | 35 (65) | 22 (50) | 30 (60)
Musculoskeletal and connective tissues (Musculoskeletal and connective tissue disorders) | 17 (20) | 14 (17) | 18 (22)
Nervous system (Nervous system disorders) | 41 (65) | 18 (31) | 28 (40)
Psychiatric (Psychiatric disorders) | 11 (12) | 10 (10) | 11 (13)
Renal and urinary (Renal and urinary disorders) | 1 (1) | 5 (10) | 8 (10)
Respiratory, thoracic and mediastinal (Respiratory, thoracic and mediastinal disorders) | 120 (385) | 65 (201) | 122 (367)
Skin and subcutaneous (Skin and subcutaneous tissue disorders) | 12 (13) | 5 (7) | 17 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT03451045/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT03451045/SAP_001.pdf